CLINICAL TRIAL: NCT06621810
Title: AI-MEL: Image Analysis and Machine Learning for Early Diagnosis and Risk Prediction in Children, Adolescents and Young Adults
Brief Title: Artificial Intelligence Based Melanoma Early Diagnosis and Risk Prediction in Children, Adolescents and Young Adults
Acronym: AI-MEL
Status: Recruiting | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: Universität Tübingen (Other); University of Florence (Other); Fundacio Clinic Barcelona (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: MELCAYA-AI-MEL
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Melanoma (Skin Cancer); Artificial Intelligence (AI); Pediatric Cancer
Keywords: melanoma; AI; pediatric; image analysis; Children Adolescence Young Adults (CAYA)
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to develop supportive diagnostic artificial intelligence algorithms to distinguish melanoma from nevi or other benign pigmented skin lesions, especially in younger patients (below the age of 30). The main goals it aims to achieve are:

* development of an algorithm based on dermatoscopic images, targeting skin cancer screening in vulnerable populations
* development of another algorithm based on histological images, intended to be used by pathologists on lesions that are still suspicious of melanoma after dermatologic assessment
* implementation of explainability methods to enable the user to better comprehend the systems' decisions, avoid biases and increase trust in these applications

There is no additional time commitment for the study participants for this study, as the data used in this project will be collected in routine clinical practice anyway.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Patients without a melanoma or nevus diagnosis
* images with insufficient image quality

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mainly children (up to and including 15 years of age), adolescents (16-20) and young adults (from 21 to 30 years of age)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operator Curve (AUROC) | First Assessment: Upon completion of the first training and testing cycle (approx. within 1.5 years from the start of the study). Reevaluations: at 6 and 12 months post-initial training for model improvement.
  The AUROC is used to measure and compare the diagnostic accuracy of different classifiers. Thereby, a higher value means better diagnostic performance, with an AUROC of 1 being a perfect score.

SECONDARY OUTCOMES:
Balanced accuracy | First Assessment: Upon completion of the first training and testing cycle (approx. within 1.5 years from the start of the study). Reevaluations: at 6 and 12 months post-initial training for model improvement.
  The balanced accuracy is used to measure and compare the diagnostic accuracy between classifier and physician. Thereby, a higher value means better diagnostic performance, with a balanced accuracy of 1 signifying perfect diagnostic capabilities.

CONTACTS AND LOCATIONS:
Overall Officials: Titus J Brinker, PD Dr. med, Principal Investigator — German Cancer Research Center
Locations (3):
- University of Tübingen, Tübingen, Germany
- University of Florence, Florence, Italy
- Hospital Clínic de Barcelona, Barcelona, Spain

REFERENCES:
- See also: Homepage of the MELCAYA project — https://melcaya.eu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT06621810/Prot_SAP_000.pdf